CLINICAL TRIAL: NCT07377409
Title: Randomised, Placebo-controlled Study to Evaluate the Beneficial Effects of Supplementation With CRONILIEF™ (Palmitoylethanolamide Phospholipids), in Addition to Standard Therapy, in Diabetic Subjects With Neuropathic Pain.
Brief Title: Beneficial Effects of Supplementation With CRONILIEF™ (Palmitoylethanolamide Phospholipids) in Diabetic Subjects With Neuropathic Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1812/28082025
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain Management; Diabetic Neuropathies, Painful; Palmitoylethanolamide
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Cronilief™ supplementation (Experimental): Cronilief™ (300 mg) supplementation
  Interventions: Dietary Supplement: Cronilief™ (300 mg)
- Group B: Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cronilief™ (300 mg) — * Week 1: Cronilief™ (300 mg), 2 tablets per day, single administration
  * Weeks 2-8: Cronilief™ (300 mg), 1 tablet per day
  Arms: Group A: Cronilief™ supplementation
Dietary Supplement: Placebo — * Week 1: Placebo, 2 tablets per day, single administration
  * Weeks 2-8: Placebo, 1 tablet per day.
  Arms: Group B: Placebo

SUMMARY:
This study aims to evaluate the potential benefit of an oral nutritional supplement based on CRONILIEF™ (Palmitoylethanolamide Phospholipids) in diabetic subjects with neuropathic pain, compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory metabolic compensation;
* Presence of moderate symptoms of painful diabetic neuropathy as assessed by the LANSS questionnaire (score ≥12);
* Taking antidiabetic drugs except insulin;
* Subjects willing and able to comply with scheduled study visits, the treatment plan, and all procedures outlined in the study.

Exclusion Criteria:

* Previous intolerance to a component of the nutraceuticals tested;
* Individuals with type I diabetes;
* Uncontrolled diabetes, severe cardiovascular and cerebrovascular diseases;
* Severe neuropathic symptoms as indicated by the LANSS score;
* Individuals undergoing insulin treatment;
* Peripheral neuropathy due to diseases other than diabetes mellitus;
* History of malignant neoplasm in the 5 years prior to enrolment in the study;
* Serious neurological, psychological or psychiatric disorders;
* Clinical signs or history of significant impairment of hepatic or renal function, peptic ulcer or coagulation disorders;
* Any clinically relevant or unstable disease (e.g., active malignancies, immune system disorders) whose sequelae or treatments could contraindicate participation in the study or interfere with the study's evaluation parameters, in the investigator's judgement; Any disease that could significantly affect the study's outcome, including, but not limited to, chronic medical conditions, psychological disorders, or substance abuse;
* Alcohol or drug abuse;
* Women of childbearing age who do not use established contraceptive methods;
* Pregnancy and breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-09-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate specific symptoms of neuropathic pain in diabetic subjects | Baseline (T0), 4 week (T1), 8 week (T2) and one month after the end of integration
  Evaluate the effectiveness of Cronilief™ supplementation versus placebo, in combination with standard therapy, in improving specific symptoms of neuropathic pain in diabetic subjects after 8 weeks of supplementation, using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) questionnaire as an assessment tool.

SECONDARY OUTCOMES:
Evaluate sleep quality | Baseline (T0), 4 week (T1), 8 week (T2) and one month after the end of integration
  Assess the impact of Cronilief™ supplementation on sleep quality, measured using the Pittsburgh Sleep Quality Index (PSQI)
Evaluate emotional states | Baseline (T0), 4 week (T1), 8 week (T2) and one month after the end of integration
  Assess the impact of Cronilief™ supplementation on emotional states related to stress, anxiety and depression through the administration of the Depression Anxiety Stress Scales (DASS-21).
Evaluate safety | Baseline (T0), 4 week (T1), 8 week (T2) and one month after the end of integration
  Assess the safety of Cronilief™ by monitoring AEs (Adverse Events) and SAEs (Serious Adverse Events) evaluated by investigators and reported in accordance with current regulations.